

Great Ormond Street London WC1N 3JH Tel: 020 7405 9200

## DEPARTMENT OF AUDIOLOGICAL MEDICINE

Consultants: Dr. E. Raglan, Dr. T. Sirimanna (Lead Clinician), Dr. K. Rajput, Dr. R. Chorbachi

(CLAP), Dr. D. Bamiou

Tel: 020 7813 8430 Fax: 020 7 829 7877

## ASSENT FORM (to be completed by children and their parents) <u>Study: FM systems on children with Auditory Processing Disorder</u> (Student Study)

## Name of researchers:

Dr. Doris-Eva Bamiou: Clinical Senior Lecturer & Consultant in Audiovestibular

Medicine

Mr. Georgios Stavrinos: PhD Student at UCL Ear Institute

Dr. Lindsey Edwards: Consultant Psychologist

Contact address: Great Ormond Street Hospital for Children NHS Trust, Great

Ormond Street, London, WC1N 3JH, Telephone: 02078138430

Please circle all the answers that you are happy with

| Have you read (or had read to you) the information about this project? | Yes / No |
|---|---|
| Do you understand what this project is about? | Yes / No |
| Do you understand it's OK to stop taking part at any time? | Yes / No |
| Are you happy to take part? | Yes / No |

| If you <u>do</u> want to take part you can write your name below.<br>Your name: |
|---|
| Your parent or carer must write their name here if they are happy for you to take part. Name of parent/carer: |
| Signature: |
| Date: |
| The researcher who explained this project to you needs to sign too. |
| Name of the person taking consent (researcher): |
| Signature: |
| Date: |